CLINICAL TRIAL: NCT00558818
Title: A Phase lV Study to Evaluate the Long-term Safety and Efficacy of Clevudine in the Patients Chronically Infected With Hepatitis B Virus
Brief Title: Long-term Study With Clevudine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: hunjun jang, Bukwang Pharmaceutical
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOR-404; KOR-404
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — clevudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clevudine — clevudine 30 mg qd

SUMMARY:
A open-labeled phase lV study with 96 weeks of treatment period. The purpose of this study is to investigate safety and efficacy of clevudine in patients chronically infected with hepatitis B virus, HBeAg positive or negative.

ELIGIBILITY:
Inclusion Criteria

* Patient with DNA levels >=1 x 10^5 copies/mL within 30 days of baseline.
* Patient is documented to be HBsAg positive for > 6 months.
* Patient has ALT levels >=80 IU/L
* Women of childbearing potential must have a negative urine (β-HCG) pregnancy test taken within 14 days of starting therapy.

Exclusion Criteria.

* Patient is currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy.
* Patients previously treated with interferon within the previous 6 months.
* Patients previously treated with clevudine, lamivudine, adefovir, entecavir, telbivudine or any other investigational nucleoside for HBV infection.
* Patient has a history of ascites, variceal hemorrhage or hepatic encephalopathy.
* Patient is coinfected with HCV, HDV or HIV.
* Patient with clinical evidence of decompensated liver disease or hepatocellular carcinoma
* Patient is pregnant or breast-feeding.
* Patient is unwilling to use an "effective" method of contraception during the study and for up to 3 months after the use of study drug ceases.
* Patient has a clinically relevant history of abuse of alcohol or drugs.
* Patient has a significant immunocompromised, gastrointestinal, renal, hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic(except HCC)or allergic disease or medical illness that in the investigator's opinion might interfere with therapy.
* Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBV DNA below the assay limit of detection by Real-time PCR | Screening, day1,every 12 weeks during treatment period(96weeks)

SECONDARY OUTCOMES:
Antiviral activity : change from baseline in HBV DNA (log10 copies/mL)Biochemical improvement (e.g. ALT normalization)Proportion of patients with HBeAg loss and/or seroconversionClevudine-related mutation | Screening, day1, every 12 weeks during treatment period(96 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- KoreaUniversity Guro Hospital, Seoul, South Korea